CLINICAL TRIAL: NCT05579665
Title: Comparative Effectiveness of Platelet Rich Plasma (PRP), Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome and Hyaluronic Acid (HA) for the Treatment of Knee Osteoarthritis
Brief Title: Effectiveness of PRP, Conditioned Medium UC-MSCs Secretome and Hyaluronic Acid for the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Collaborators: Dr. Mohammad Hoesin Central General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58/kepkrsmh/2022
Record Dates: First submitted 2022-10-04; First posted 2022-10-14 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Secretome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet-rich Plasma (PRP) (Experimental): Platelet-rich plasma administered 5 times as an intra-articular injection under ultrasound guidance as a series of one weekly injections to the affected knee. 1 weekly injections are of leukocyte poor, buffer/additive free, singe spin, platelet-rich plasma averaging 3mL in volume.
  Interventions: Biological: Platelet-rich Plasma
- Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome (Experimental): Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome administered 5 times as an intra-articular injection under ultrasound guidance as a series of one weekly injections to the affected knee. 1 weekly injections are Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome averaging 2 mL in volume.
  Interventions: Biological: Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome
- Hyaluronic Acid (HA) (Experimental): Hyaluronic Acid administered 5 times as an intra-articular injection under ultrasound guidance as a series of one weekly injections to the affected knee. 1 weekly injections are of low molecular weight hyaluronan in a 2mL injection.
  Interventions: Drug: Low Molecular Weight Hyaluronic Acid

INTERVENTIONS:
Biological: Platelet-rich Plasma — Research participants own blood will be used to prepare the platelet rich plasma injectate.
  Other Names: PRP
  Arms: Platelet-rich Plasma (PRP)
Biological: Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome — Conditioned Medium UC-MSCs Secretome which will be injected into the affected knee using ultrasound guidance.
  Other Names: Conditioned Medium UC-MSCs Secretome
  Arms: Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell Culture (MSCs) Secretome
Drug: Low Molecular Weight Hyaluronic Acid — low molecular weight hyaluronic acid which will be injected into the affected knee using ultrasound guidance.
  Other Names: HA
  Arms: Hyaluronic Acid (HA)

SUMMARY:
The clinical trial will be carried out at the Dr. Moh. Hoesin Central Hospital, Palembang and planned from October 2022 to March 2023.

This study aims to compare the efficacy of Platelet Rich Plasma, Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell (MSC) Culture Secretome and hyaluronic acid for the Treatment of Knee Osteoarthritis

DETAILED DESCRIPTION:
In this, prospective, Open-label study, patients with mild to moderate symptomatic knee osteoarthritis will be randomized to receive either a series of platelet-rich plasma or hyaluronic acid or Conditioned Medium From Umbilical Cord Mesenchymal Stem Cell (MSC) Culture Secretome injections under ultrasound guidance. Each of the groups were given 5 times injection 3 cc platelet-rich plasma or 2 cc hyaluronic acid or 2cc Conditioned Medium From Umbilical Cord MSC Secretome at intervals 1 weeks.

Clinical data in the form of subjective outcome measures will be collected pre-treatment and 6 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-60 years
* Suffering from grade 2 and 3 osteoarthritis (OA) was identified by two observers who differed accordingly the Kellgren and Lawrence research scale
* Patient with knee pain that had been continuing for at least 12 months with no relief using anti-inﬂammatory medications and that deteriorated with weight-bearing
* Patients can understand the nature of the study and written informed consent is given to patients

Exclusion Criteria:

* Age > 60 years
* Acute Knee Osteoarthritis Effusions
* Patients are not willing to obey the study protocol
* There are signs of infection local or general infection or positive serology for HIV, hepatitis and syphilis
* There is a congenital disease that causes significant deformity of the knee can interfere with cell applications and interpret results
* Articular injection of the knee by any drug during the previous 3 months
* Participate in any clinical trial or treatment 30 days before the study
* Other conditions may, according to medical criteria, not support participation in this research (The recent history of knee trauma, Autoimmune rheumatic diseases, Uncontrolled systemic diseases such as diabetes or hypertension, patient with Immunosuppressive or anticoagulant treatment and cancer)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Pre-Treatment
  To asses pain score, score 1(good)-10(worst)
Visual Analog Scale (VAS) | 3 month after injection
  To asses pain score, score 1(good)-10(worst)
Visual Analog Scale (VAS) | 6 month after injection
  To asses pain score, score 1(good)-10(worst)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Pre-Treatment
  To evaluate the condition of patients with osteoarthritis, including pain, stiffness, and physical functioning of the joints. The WOMAC is a self administered questionnaire consisting of 24 items divided into subscales including pain (0-20), stiffness (0-8) and physical function (0-68). Higher scores indicate worse pain, stiffness and functional limitations.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 month after injection
  To evaluate the condition of patients with osteoarthritis, including pain, stiffness, and physical functioning of the joints. The WOMAC is a self administered questionnaire consisting of 24 items divided into subscales including pain (0-20), stiffness (0-8) and physical function (0-68). Higher scores indicate worse pain, stiffness and functional limitations.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 month after injection
  To evaluate the condition of patients with osteoarthritis, including pain, stiffness, and physical functioning of the joints. The WOMAC is a self administered questionnaire consisting of 24 items divided into subscales including pain (0-20), stiffness (0-8) and physical function (0-68). Higher scores indicate worse pain, stiffness and functional limitations.

SECONDARY OUTCOMES:
Laboratory Assessment | Pre-Treatment
  Cartilage Oligomeric Matrix Protein (COMP)
Laboratory Assessment | 3 month after injection
  Cartilage Oligomeric Matrix Protein (COMP)

CONTACTS AND LOCATIONS:
Overall Officials: Radiyati U Partan, MD, Principal Investigator — Universitas Sriwijaya; Surya Darma, MD, Study Director — Universitas Sriwijaya
Locations (1):
- Mohammad Hoesin Central General HospitalPalembang, Palembang, South Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerza F, Carni S, Carcangiu A, Di Vavo I, Schiavilla V, Pecora A, De Biasi G, Ciuffreda M. Comparison between hyaluronic acid and platelet-rich plasma, intra-articular infiltration in the treatment of gonarthrosis. Am J Sports Med. 2012 Dec;40(12):2822-7. doi: 10.1177/0363546512461902. Epub 2012 Oct 25. PMID 23104611
- [Background] Raeissadat SA, Rayegani SM, Hassanabadi H, Fathi M, Ghorbani E, Babaee M, Azma K. Knee Osteoarthritis Injection Choices: Platelet- Rich Plasma (PRP) Versus Hyaluronic Acid (A one-year randomized clinical trial). Clin Med Insights Arthritis Musculoskelet Disord. 2015 Jan 7;8:1-8. doi: 10.4137/CMAMD.S17894. eCollection 2015. PMID 25624776
- [Background] Montanez-Heredia E, Irizar S, Huertas PJ, Otero E, Del Valle M, Prat I, Diaz-Gallardo MS, Peran M, Marchal JA, Hernandez-Lamas Mdel C. Intra-Articular Injections of Platelet-Rich Plasma versus Hyaluronic Acid in the Treatment of Osteoarthritic Knee Pain: A Randomized Clinical Trial in the Context of the Spanish National Health Care System. Int J Mol Sci. 2016 Jul 2;17(7):1064. doi: 10.3390/ijms17071064. PMID 27384560
- [Background] Magnussen RA, Flanigan DC, Pedroza AD, Heinlein KA, Kaeding CC. Platelet rich plasma use in allograft ACL reconstructions: two-year clinical results of a MOON cohort study. Knee. 2013 Aug;20(4):277-80. doi: 10.1016/j.knee.2012.12.001. Epub 2012 Dec 24. PMID 23270598
- [Background] Ossendorff R, Walter SG, Schildberg FA, Khoury M, Salzmann GM. Controversies in regenerative medicine: should knee joint osteoarthritis be treated with mesenchymal stromal cells? Eur Cell Mater. 2022 Mar 17;43:98-111. doi: 10.22203/eCM.v043a09. PMID 35298024
- [Background] Gosens T, Den Oudsten BL, Fievez E, van 't Spijker P, Fievez A. Pain and activity levels before and after platelet-rich plasma injection treatment of patellar tendinopathy: a prospective cohort study and the influence of previous treatments. Int Orthop. 2012 Sep;36(9):1941-6. doi: 10.1007/s00264-012-1540-7. Epub 2012 Apr 27. PMID 22534958

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT05579665/Prot_ICF_000.pdf